CLINICAL TRIAL: NCT04352868
Title: Customizing Myopia Control With Multifocal Toric Contact Lens
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Andrew Pucker, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300004596
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Refractive Errors; Myopia
Keywords: Myopia; Multifocal contact lens; Refractive error; Myopia treatment; Myopia control; Myopia management
MeSH Terms: conditions — Refractive Errors; Myopia | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Toric soft contact lens (Active Comparator): Toric soft contact lens
  Interventions: Device: Intelliwave toric, soft contact lens
- Multifocal toric soft contact lens (Experimental): A multifocal toric soft contact lens with a +2.00 D add.
  Interventions: Device: Intelliwave multifocal, toric, soft contact lens

INTERVENTIONS:
Device: Intelliwave multifocal, toric, soft contact lens — This is a quarterly disposable, multifocal, toric soft contact lens commercially available from Art Optical Contact Lens, Inc.
  Arms: Multifocal toric soft contact lens
Device: Intelliwave toric, soft contact lens — This is a quarterly disposable toric soft contact lens commercially available from Art Optical Contact Lens, Inc.
  Arms: Toric soft contact lens

SUMMARY:
This study will evaluate the ability of toric multifocal contact lens to reduce the change of myopia progression in children (aged 8-12) with myopic astigmatism.

DETAILED DESCRIPTION:
The purpose of this study is to assess if a center distance toric multifocal contact lenses can slow the amount of change of myopia progression in children with myopia plus astigmatism. Multifocal contact lenses have been theorized to influence the peripheral optics of the eye such that they slow the rate of myopia progression in nearsighted children. This outcome is yet to be evaluated in children with myopia plus astigmatism.The secondary outcome is to measure the change in peripheral optics caused by the contact lens. This information is key to understanding the mechanism of multifocal contact lens optics on the eye. Ultimately this information would be used to create a software that can estimate the effect of multifocal contact lenses on the peripheral optics of the child's eye. This software can potentially be used by practitioners worldwide to better customize multifocal contact lenses to slow myopia progression.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 12 years, inclusive, at baseline examination
* -0.50 to -6.00 D, inclusive, spherical component, cycloplegic autorefraction
* ≥0.75 DC, cycloplegic autorefraction
* 0.1 logMAR or better best-corrected visual acuity in each eye

Exclusion Criteria:

* Eye disease or refractive error conditions (e.g., keratoconus, retinal abnormalities, retinopathy of prematurity, etc.)
* Ocular surgery, severe ocular trauma, active ocular infection or inflammation
* Subjects with a condition or in a situation, which in the examiner's opinion, may put the subject at significant risk, may confound the study results, or may significantly interfere with their participation in the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Refractive error progression | 1 years
  Refractive error measured by cycloplegic autorefraction in both eyes, will be measured at baseline and at one year to assess the difference in spherical component of the refractive error between the treatment group (multifocal toric soft contact lens) and the control group (toric soft contact lens)
Axial length | 1 years
  Change in axial length as measured by non-contact axial length both eyes, will be measured at baseline and at one year to assess the difference in change in axial length between the treatment group (multifocal toric soft contact lens) and the control group (toric soft contact lens)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Pucker, OD, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual subject data.